CLINICAL TRIAL: NCT04506983
Title: The Phase I Efficacy and Safety Clinical Study of GPC3-CAR-T Cells in Hepatocellular Carcinoma Patients
Brief Title: GPC3-CAR-T Cells for the Hepatocellular Carcinoma
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Adjust the plan
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Collaborators: China Immunotech (Beijing) Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HXYT-009
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GPC3-CAR-T cells (Experimental): Patients with hepatocellular carcinoma will be enrolled, and GPC3-CAR-T cells will be intravenously infused with a escalated dose of 1×106 /3×106/10×106GPC3-CAR-T cells. Tumor markers and GPC3-CAR-T cell proliferation will be monitored in the scheduled time (day 0, day 4, day 7, day 10, day 14,day 21, day 28).
  Interventions: Biological: GPC3-CAR-T cells

INTERVENTIONS:
Biological: GPC3-CAR-T cells — Patients with hepatocellular carcinoma will be enrolled, and GPC3-CAR-T cells will be intravenously infused with a escalated dose of 1×106 /3×106/10×106GPC3-CAR-T cells.

SUMMARY:
This is a single center, single arm, open-label, phase I study to evaluate the safety and efficacy of GPC3-CAR-T cells in patients with hepatocellular carcinoma.

DETAILED DESCRIPTION:
GPC3-CAR-T cells is a novel CAR-T cells which designed for the cell membrane protein Glypican-3. Patients with hepatocellular carcinoma will be enrolled, and GPC3-CAR-T cells will be intravenously infused with a escalated dose of 1×106, 3×106, 10×106 GPC3-CAR-T cells. Tumor markers and GPC3-CAR-T cell proliferation will be monitored in the scheduled time (day 0, day 4, day 7, day 10, day 14, day 28). The aim of this clinical trial is to evaluate the safety and efficacy of GPC3-CAR-T cells therapy in patients with hepatocellular carcinoma. The primary endpoint is the safety of CAR-T cells including the effect ratio of CRS and ICANS, ORR. The secondary endpoint is the CAR-T ratio and CAR gene copied number in PB, PFS, OS and DOR.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≧18years, gender unlimited.
2. Failure or intolerance after at least first-line treatment.
3. GPC3 positive(IHC)
4. Patients must have at least one target lesion available for evaluation.
5. BCLC B or C.
6. Child-Pugh grade A or B
7. ECOG is 0 or 1 (one week before enrollment.)
8. Estimated life expectancy ≥ 3 months.
9. Functioning of major organs are normal.
10. Women of childbearing age (15-49 years old) must receive a pregnancy test within 7 days prior to initiation of treatment and the results are negative; male and female patients with fertility must use an effective contraceptive to ensure 3 months after discontinuation of treatment during the study period not pregnant inside.
11. Patients who voluntarily sign informed consent and are willing to comply with treatment plans, visit arrangements, laboratory tests and other research procedures.

Exclusion Criteria:

1. There are uncontrollable active infections that need systemic treatment.
2. HIV antibody is positive or syphilis antibody is positive.
3. Pregnant or lactating women.
4. hepatic encephalopathy.
5. patients with organ failure:

   * Heart: NYHA heart function grade IV;
   * Liver: Grade C that achieves Child-Turcotte liver function grading;
   * Kidney: kidney failure and uremia;
   * Lung: symptoms of respiratory failure;
   * Brain: a person with a disability.
6. It is undergoing systemic hormones therapy.
7. Impact results show that over 50% of the liver is occupied by tumor .
8. Patients who are still in the observation stage of other antitumor drugs 30 days before blood collection.
9. Patients were received other gene therapy products, or are participating in other clinical trials within 4 weeks prior to cell infusion.
10. Abnormal thyroid function ≧Level 3.
11. Active autoimmune diseases require systemic treatment during the first two years of screening.
12. Patients have mental illness or history of drug abuse.
13. Patients are participating in other clinical studies.
14. The researchers found that it was unsuitable for the recipients to be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-06-10 (Estimated); Primary Completion 2023-06-10 (Estimated); Study Completion 2023-10-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of adverse events | 12months
  Percentage of participants with adverse events.

SECONDARY OUTCOMES:
Objective Remission Rate(ORR) | 12months
  The percentage of participants who achieved complete remission (CR) and partial remission over all participants.
Proliferation ratio of CAR-T cells | 12months

CONTACTS AND LOCATIONS:
Overall Officials: Gong Li, M.A., Study Director — Beijing Tsinghua Changgeng Hospital
Locations (1):
- Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality, China